CLINICAL TRIAL: NCT02238327
Title: The Study is a Multicenter, Prospective Observational Study of Pathogenesis of HIV Pulmonary Disease.
Brief Title: Longitudinal Evaluation of HIV-associated Lung Disease Phenotypes
Acronym: LEAP
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alison Morris, Professor, University of Pittsburgh
Other Study IDs: PRO14070355; 1R01HL125049-01 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; HIV; Emphysema
Keywords: Antiretroviral therapy; pulmonary function; biomarkers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Blood Specimen Collection; Surveys and Questionnaires; Nasal Lavage; Caves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, bronchial wash and cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV positive normal pulmonary function: HIV positive DLCO percent predicted >=.80 FEV1/FVC percent predicted >=0.70
  Interventions: Procedure: blood draw; Procedure: questionnaires; Procedure: Lung function testing; Procedure: Six-Minute walk test; Radiation: Quantitative CT scans; Procedure: Nasal secretion and cell collection; Procedure: Echocardiogram
- HIV positive with pulmonary dysfuntion: HIV positive DLco percent predicted <=0.80% FEV1/FVC percent predicted<=0.70%
  Interventions: Procedure: blood draw; Procedure: questionnaires; Procedure: Lung function testing; Procedure: Six-Minute walk test; Radiation: Quantitative CT scans; Procedure: Nasal secretion and cell collection; Procedure: Echocardiogram

INTERVENTIONS:
Procedure: blood draw — Blood will be drawn for plasma, serum, and PBMCs. Clinical labs drawn will be for hepatitis, CMV, hemoglobin and carboxyhemoglobin.
Procedure: questionnaires — The following questionnaires are administered to participants by study personnel at each visit: LEAP questionnaire, St. George's, and MMRC.
Procedure: Lung function testing — The routine lung function endpoints of FVC, FEV1, FEV1/FVC, and FEF25-75% will be measured before and after bronchodilator administration (4 puffs of albuterol). The best of three reproducible forced expiratory attempts is used in analysis. Percent- predicted spirometric values are based on age, height, gender, and ethnicity. DLco will be measured using the automated single-breath procedure of the integrated testing system, which conforms to ATS standards. DLco will be adjusted for hemoglobin and carboxyhemoglobin.
  Other Names: Spirometry
Procedure: Six-Minute walk test — Six-minute walk tests are performed in a 100 foot (30.48 m) segment of straight hallway marked at 10 foot (3 m) intervals. In addition to the usual ATS protocol, the patient is monitored, when available, with Bluetooth wireless pulse oximetry and the time and distance recorded after six minutes and if they desaturate to <88%. Dyspnea (Borg 0-10) and perceived exertion (Borg 6-20) scales are completed at the beginning and the end of test.
Radiation: Quantitative CT scans — Subjects will undergo a standard chest CT. The CT scans will use a phantom shipped between sites to standardize results and capture contiguous volume scans acquired at slice thicknesses of 5.0 mm in the axial plane and reconstructed with 512 x 512 pixel matrices. CT examinations will encompass the entire thorax and be performed during a breath-hold at end-inspiration. We will measure % of lung tissue below a threshold for emphysema (i.e. -950 Hounsfield units). Measurements have been histologically-verified and give reproducible measurements. The data set is assembled and analyzed with the image data anonymized.
  Other Names: CT scan of the chest
Procedure: Nasal secretion and cell collection — Participants will be instructed to blow their nose to remove accumulated mucus. Two sprays of commercially available nasal saline will be instilled in each nostril. The participant will then be ask to exhale through the rinsed nostril into a specimen cup. We will repeat this up to 5 times on each side depending on the participants' tolerance to the procedure. Using an otoscope, a small curette will then be used to collect 3 to 5 samples of nasal cells from each nostril. These samples will be used immediately for analysis or banked for future study.
  Other Names: Nasal wash; Nasal scrapping
Procedure: Echocardiogram — The cardiac ultrasound will use standard ultrasound techniques to image two-dimensional slices of the heart using 3D real-time imaging.
  Other Names: Echo

SUMMARY:
The overall hypotheses of this proposal are that discrete phenotypes of HIV Chronic Obstructive Pulmonary disease (COPD) differ in their trajectories, biomarkers, and risk factors and that persistent viral infection including residual HIV is linked to HIV COPD.

DETAILED DESCRIPTION:
The study is a multicenter, prospective observational study of pathogenesis of HIV pulmonary disease. We will determine the prevalence and risk factors for lung dysfunction as quantified by pulmonary function testing in HIV+ subjects. We will build on our existing longitudinal cohorts while adjusting for important co-variates such as antiretroviral therapy (ART), smoking history, co-infections, and illicit drug use. Evaluations will be scheduled at baseline, 18 months, and 36 months. (6, 12, 18 and 36 months for ART initiators at the UCSF). Study visits will consist of blood draw, questionnaires, pulmonary function testing, 6-minute walk test, CT of the chest at visit two. Oral specimen collection and glycocalyx and echocardiogram (visit two) at the Pittsburgh site only.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented in medical record at any time prior to study entry.
* Men and women age 18 to 80.
* Ability and willingness to complete all tests.
* Participant in HLRC studies, MACS, Women's Interagency Health Study, and local HIV clinics.
* For UCSF only, new ART initiators from Women's Interagency Health Study or the HIV clinic

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Contraindication to pulmonary function testing (i.e. abdominal or cataract surgery within 3 months, recent myocardial infarction, etc.).
* Increasing respiratory symptoms or febrile (temperature >100.40F [380C]) within 4 weeks of study entry.
* Hospitalization within 4 weeks prior to study entry (excluding mental health).
* Uncontrolled hypertension at screening visit (systolic > 180 mm Hg or diastolic > 100 mm Hg) from an average of two or more readings. Subject may return for screening after blood pressure is controlled.
* Active cancer requiring systemic chemotherapy or radiation.
* Active infection of lungs, brain, or abdomen.
* Intravenous drug use or alcohol use that will impair ability to complete study investigations in the opinion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be HIV positive subjects previously seen for other studies. There will be three centers enrolling, the University of Pittsburgh, the University of California San Francisco, and the University of California Los Angeles. Recruitment will occur from participants in ongoing lung studies at these sites.
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
differences in the trajectory of FEV1 in clinical COPD phenotypes, | 36 months
  PFT's at baseline, 18 months and 36months to determine modifying risk factors and relationship of phenotypes to mortality, and delineate the association of ART and lung dysfunction.

SECONDARY OUTCOMES:
will measure biomarkers of these phenotypes and ability to predict HIV COPD | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Drummond MB, Huang L, Diaz PT, Kirk GD, Kleerup EC, Morris A, Rom W, Weiden MD, Zhao E, Thompson B, Crothers K. Factors associated with abnormal spirometry among HIV-infected individuals. AIDS. 2015 Aug 24;29(13):1691-700. doi: 10.1097/QAD.0000000000000750. PMID 26372280
- [Background] Gingo MR, Nouraie M, Kessinger CJ, Greenblatt RM, Huang L, Kleerup EC, Kingsley L, McMahon DK, Morris A. Decreased Lung Function and All-Cause Mortality in HIV-infected Individuals. Ann Am Thorac Soc. 2018 Feb;15(2):192-199. doi: 10.1513/AnnalsATS.201606-492OC. PMID 29313714
- [Background] Qin S, Clausen E, Nouraie SM, Kingsley L, McMahon D, Kleerup E, Huang L, Ghedin E, Greenblatt RM, Morris A. Tropheryma whipplei colonization in HIV-infected individuals is not associated with lung function or inflammation. PLoS One. 2018 Oct 4;13(10):e0205065. doi: 10.1371/journal.pone.0205065. eCollection 2018. PMID 30286195